CLINICAL TRIAL: NCT07068126
Title: "The Safety and Efficacy of Mini-Pool IVIG Initiation and Maintenance Therapy for Management of Children With Persistent ITP, A Novel Approach for LMICs"
Brief Title: Management of Children With Persistent ITP, A Novel Approach
Acronym: LMICs
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Collaborators: Zagazig University (Other Government); Ain Shams University (Other)
Responsible Party: Principal Investigator, Mervat A. M. Youssef, Principal investigator, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB:04-2025-300549; IRB:04-2025-300549 (Other: Assuit University)
Record Dates: First submitted 2025-07-02; First posted 2025-07-16 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Persistent Immune Thrombocytopenia

STUDY DESIGN:
Intervention Model Description: All enrolled participants will receive mini-pool intravenous immunoglobulin (IVIG) as a second-line treatment for persistent immune thrombocytopenia (ITP). The study follows a single-group assignment model with no control or comparison group. Dosing intervals are adjusted based on each participant's platelet count response.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Mini-Pool IVIG Treatment Arm (Experimental): Participants in this arm will receive mini-pool intravenous immunoglobulin (IVIG) as second-line therapy for persistent immune thrombocytopenia (ITP). Treatment includes a loading dose of 1 g/kg infused over 6-8 hours, followed by maintenance doses of 0.5 g/kg given every 2 to 4 weeks for up to five additional doses. The dosing interval is adjusted based on each participant's platelet count. Participants will have regular blood tests and clinical assessments to monitor platelet levels, bleeding episodes, and treatment safety.
  Interventions: Biological: Mini-Pool IVIG

INTERVENTIONS:
Biological: Mini-Pool IVIG — Mini-pool intravenous immunoglobulin (IVIG) is a plasma-derived biologic prepared from small pools of locally donated human plasma using a validated, virus-inactivated, closed-system process. Each participant will receive a loading dose of 1 g/kg infused intravenously over 6-8 hours. Maintenance doses of 0.5 g/kg will be given every 2 to 4 weeks for up to five additional doses, with the dosing schedule adjusted based on platelet count. The preparation contains purified IgG and meets safety standards for sterility and viral inactivation.

SUMMARY:
The goal of this clinical trial is to learn if mini-pool intravenous immunoglobulin (IVIG) is a safe and effective treatment for children with persistent immune thrombocytopenia (ITP). ITP is a condition that causes low platelet levels and increases the risk of bleeding. The main questions this study aims to answer are:

Can mini-pool IVIG raise platelet levels in children with persistent ITP?

Can it reduce bleeding episodes and hospital visits?

What side effects, if any, are seen with this treatment?

There is no comparison group in this study. All participants will receive mini-pool IVIG, which is made from small pools of donated plasma using a cost-effective process.

Participants will:

Receive one dose of mini-pool IVIG through a vein over 6 to 8 hours

Receive follow-up doses every 2 to 4 weeks for up to 5 doses, based on their platelet count

Have regular blood tests and checkups during the study and for 6 months after treatment

Report on bleeding episodes, physical activity, school attendance, and side effects

DETAILED DESCRIPTION:
Immune thrombocytopenia (ITP) is an autoimmune condition where the immune system destroys platelets, leading to low platelet counts and increased risk of bleeding. Persistent ITP is defined as ongoing thrombocytopenia lasting 3 to 12 months after initial diagnosis. Children with persistent ITP who lose their response to first-line treatments, such as steroids or standard intravenous immunoglobulin (IVIG), have limited therapeutic options, especially in low- and middle-income countries, due to the high cost of commercial IVIG preparations.

Mini-pool IVIG is produced from small pools of plasma collected locally, using a validated process with virus inactivation and IgG purification steps. This method enables safe, cost-effective preparation of IVIG in resource-limited settings. Prior research has shown that mini-pool IVIG is effective and well-tolerated in acute pediatric ITP, but its role as a second-line therapy for persistent ITP has not been evaluated.

This multicenter, prospective clinical trial will enroll 20 children aged 1 to 10 years with persistent ITP at three tertiary care pediatric hematology centers in Egypt. Participants will receive a loading dose of mini-pool IVIG at 1 g/kg, followed by maintenance doses of 0.5 g/kg every 2 to 4 weeks for up to five additional doses, with dose intervals adjusted based on platelet counts.

Throughout the study, participants will undergo regular blood counts, bleeding assessments using the Bleeding Assessment Tool (BAT), and monitoring for infusion-related or delayed adverse events. Data on school attendance, physical activity, and patient or family satisfaction will also be collected.

Responses to therapy will be classified as complete response (CR), response (R), or no response (NR) based on platelet count thresholds and bleeding status, with response duration measured from achievement of CR or R to loss of response. Participants achieving sustained response off therapy (SRoT) or response off therapy (RoT) during the 6-month post-treatment follow-up will be identified to evaluate durability of treatment effects.

This study aims to provide evidence on the safety and efficacy of mini-pool IVIG as a second-line therapy for persistent pediatric ITP, potentially offering an affordable and effective treatment alternative in settings where standard IVIG is inaccessible due to cost.

ELIGIBILITY:
Inclusion Criteria:Age 1 - 10 years

* Gender: Males and Females
* Persistent ITP according to ASH definition
* No history of treatment with thrombopoietin agonists

Exclusion Criteria:-History of severe drug adverse events to IVIG

* Previous history of ICH
* Difficult venous access
* Congenital thrombocytopenia, secondary ITP and non-immune thrombocytopenia

Ages: 1 Year to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Bleeding Frequency and Severity | From enrollment through 6 months post-treatment.
  Number, location, and severity of bleeding episodes assessed using the Bleeding assessed using the ISTH Bleeding Assessment Tool (BAT) score, which evaluates bleeding symptoms across multiple anatomical sites. Each site is scored from 0 to 4, with higher scores indicating more severe bleeding. The total score varies depending on the number and severity of bleeding events.Assessment Tool (BAT) score.
Platelet Count Response | Assessed monthly during treatment and for 6 months after last dose.
  Number of participants achieving complete response (platelet count ≥100×10⁹/L) or response (platelet count ≥30×10⁹/L and at least 2-fold increase from baseline) without bleeding.
Frequency of Hospital Admissions Due to Critical Bleeding | From enrollment through 6 months post-treatment.
  Number of hospital admissions for life-threatening bleeding episodes, excluding admissions solely for IVIG infusion.

SECONDARY OUTCOMES:
Adverse Events | From first infusion through 6 months after the last dose.
  Number and type of infusion-related or delayed adverse events experienced during or after mini-pool IVIG treatment.
School Attendance | From enrollment through 6 months post-treatment.
  Change in days missed from school compared to baseline, as a measure of quality of life.
Patient and Family Satisfaction | Assessed at the end of treatment and at 6-month follow-up.
  Level of satisfaction with mini-pool IVIG treatment as reported by participants and caregivers using a structured satisfaction questionnaire.
Sustained Response Off-Therapy (SRoT/RoT) | 6 months after last mini-pool IVIG dose.
  number of participants maintaining platelet counts ≥100×10⁹/L (SRoT) or ≥30×10⁹/L without bleeding (RoT) for at least 6 months after completing mini-pool IVIG therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Mervat M A Youssef, Assistant Professor, Principal Investigator — Assiut University
Locations (3):
- Egypt (3):
  - Children's hospital - Assiut University, Asyut
  - Ain Shams University, Cairo
  - Zagazig University, Pediatric departement, Zagazig

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] 1. Kohli, R. and S. Chaturvedi, Epidemiology and Clinical Manifestations of Immune Thrombocytopenia. Hamostaseologie, 2019. 39(3): p. 238-249. 2. Pietras, N.M., et al., Immune Thrombocytopenia, in StatPearls. 2024, StatPearls Publishing Copyright © 2024, StatPearls Publishing LLC.: Treasure Island (FL). 3. Thakur, Y., R.J. Meshram, and A. Taksande, Diagnosis and Management of Immune Thrombocytopenia in Paediatrics: A Comprehensive Review. Cureus, 2024. 16(9): p. e69635. 4. Wang, Z., et al., Sustained response off treatment in eltrombopag for children with persistent/chronic primary immune thrombocytopenia: A multicentre observational retrospective study in China. Br J Haematol, 2023. 202(2): p. 422-428. 5. Gotesman, M., et al., Pediatric Immune Thrombocytopenia. Adv Pediatr, 2024. 71(1): p. 229-240. 6. El-Ekiaby, M., et al., Minipool caprylic acid fractionation of plasma using disposable equipment: a practical method to enhance immunoglobulin supply in developing countries. PLoS Negl Trop Dis, 2015. 9(2): p. e0003501. 7. Elalfy, M., et al., A randomized multicenter study: safety and efficacy of mini-pool intravenous immunoglobulin versus standard immunoglobulin in children aged 1-18 years with immune thrombocytopenia. Transfusion, 2017. 57(12): p. 3019-3025. 8. Rodeghiero, F., et al., Standardization of terminology, definitions and outcome criteria in immune thrombocytopenic purpura of adults and children: report from an international working group. Blood, 2009. 113(11): p. 2386-93.

DOCUMENTS (1):
  • Study Protocol (2024-12-24): https://cdn.clinicaltrials.gov/large-docs/26/NCT07068126/Prot_000.pdf